CLINICAL TRIAL: NCT07295990
Title: The Impact of Dysphagia Exercise on Oropharyngeal Swallowing Function in Patients With ALS
Brief Title: Tongue-strengthening Exercises in People With ALS.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dysphagia Exercise ALS
Record Dates: First submitted 2025-12-03; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: ALS (Amyotrophic Lateral Sclerosis); ALS - Amyotrophic Lateral Sclerosis
Keywords: ALS; Amyotrophic Lateral Sclerosis; Dysphagia; Dysarthria
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Deglutition Disorders; Dysarthria

STUDY DESIGN:
Intervention Model Description: Delayed start, repeated-measures design,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dysphagia Exercise Intervention (Experimental): This study arm will test a proactive dysphagia exercise program using lingual manometry and isometric lingual strength training in people with ALS (pALS). The intervention is designed to maximize lingual strength, improve speech intelligibility, enhance swallow safety and efficiency, and support patient-reported swallowing and quality-of-life outcomes in individuals with minimal decline in tongue function.
  Interventions: Procedure: Isometric Lingual Strength Exercises

INTERVENTIONS:
Procedure: Isometric Lingual Strength Exercises — Direct intervention will consist of an isometric lingual exercise program designed specifically for patients with ALS. Participants will complete five exercise sessions per week for a total of five weeks, with each session including six sets of five repetitions (30 repetitions daily, 150 repetitions weekly). Exercises will be performed at 60% of each participant's maximum isometric anterior lingual pressure (MAIP), with each tongue press held for approximately two seconds. Training thresholds will be adjusted weekly via telehealth to ensure the program remains at the prescribed 60% intensity, supporting both safety and consistency in progression. This structured protocol is intended to maximize lingual strength, swallow function, and overall adherence to the intervention.

SUMMARY:
This study is testing a tongue exercise program for people living with ALS to see if it can help support speech and swallowing. All participants will receive the treatment, and researchers will measure changes over time by comparing each person's results to their own earlier results.

People who join the study will have two in-person visits, one virtual visit, and four weekly telehealth sessions with a speech-language pathologist. During these sessions, participants will practice tongue resistance exercises, complete speech and swallowing tasks, and answer surveys about their experience. They will also use a small device at home to measure tongue strength and swallowing.

The exercise program involves pressing the tongue against a device several times a day, five days per week, for five weeks. Researchers want to learn if this program is safe, practical, and helpful for people with ALS.

DETAILED DESCRIPTION:
Study Description

Brief Summary:

This study is designed to evaluate the effects of isometric lingual strengthening exercises on speech and swallowing function in individuals with Amyotrophic Lateral Sclerosis (ALS). By targeting tongue strength, we aim to improve pressure generation, support safer and more efficient swallowing, enhance speech intelligibility, and examine the relationship between lingual strength and patient-reported outcomes.

Detailed Description:

Amyotrophic Lateral Sclerosis (ALS) often results in progressive weakness of the tongue and other oral structures, which contributes to impaired speech intelligibility, swallowing safety, and overall quality of life. Lingual strengthening exercises may offer a non-invasive, behavioral intervention to preserve oral function in this population. However, the efficacy and broader impact of such exercises remain underexplored.

The aims of this study are to:

Evaluate the efficacy of isometric lingual strength exercises in improving tongue pressure generation in people with ALS (pALS).

Investigate the impact of lingual strengthening exercises on speech intelligibility, swallowing safety, and swallowing efficiency.

Assess the relationship between lingual strength, speech intelligibility, swallowing function, and patient-reported outcomes related to motor speech, swallowing-related quality of life, and fatigue.

Methods and Study Design:

This study uses a delayed-start, repeated-measures design in which participants serve as their own controls. This approach allows all participants to receive the intervention while also accounting for disease heterogeneity and interparticipant variability.

Participants will complete two baseline assessments (in-person at Week 0, virtual at Week 5), a 5-week intervention phase (Weeks 5-10), and a final in-person evaluation at Week 10. A follow-up strength assessment will occur at the participant's next scheduled multidisciplinary ALS Clinic visit (~6 months).

Study Procedures and Timeline:

Screening / Baseline 1 (Week 0, in-person, 60-90 min):

Informed consent and eligibility screening.

Assessments: Maximum isometric lingual pressure (Tongueometer), 3D tongue ultrasound, Bamboo Passage (speech rate), oral diadochokinesis (temporal variability), 3-ounce water test (swallowing safety), TOMASS (oral efficiency), videofluoroscopic swallow study (VFSS), and patient-reported measures (Eat-10, ALSFRS-R, ETBQ).

Baseline 2 (Week 5, virtual, 60-90 min):

Repeat assessments from Baseline 1, excluding VFSS and ultrasound.

Introduction of isometric lingual strength training; first training session completed during this visit.

Telehealth Training Sessions (Weeks 5-10, weekly, 30-60 min each):

Conducted via Zoom.

Tongue resistance training, Bamboo Passage, diadochokinesis, 3-ounce water test.

Patient-reported measures (ALSFRS-R, ETBQ, Eat-10).

Research clinician monitors fidelity, provides progression adjustments, and records data.

Active Exercise Training Regimen:

Frequency: 5 sessions per week for 5 weeks.

Intensity: 60% of each participant's maximum anterior lingual pressure (MAIP).

Volume: 6 sets of 5 repetitions/day (30 repetitions/day; 150 repetitions/week).

Contraction: 2-second hold for each isometric press.

Progression: Training thresholds updated weekly to maintain 60% MAIP.

Final Evaluation (Week 10, in-person):

Assessments identical to Baseline 2 with inclusion of VFSS, ultrasound, and ETBQ.

Follow-up (6 months, routine ALS clinic visit):

Isometric lingual strength assessment repeated using the Tongueometer.

Exploratory Outcome:

Ultrasound imaging will be completed at baseline and final evaluations to quantify morphologic changes in tongue structure related to exercise.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of possible, probable, or definite ALS (El-Escorial Revisited)
* Lingual exercises naïve
* Impaired lingual strength generation compared to normative data (<43 kPa; Robinson et al., 2023)
* EAT-10 score <3

Exclusion Criteria:

* Stroke
* Head injury
* Head and neck cancer
* Tracheostomy
* Other concomitant neurogenic disorder
* Recent oral surgery other than routine dental surgery
* Unable to generate isometric lingual pressure on lingual manometer
* Participation in another clinical trial intervention that may confound results
* NPO (nothing by mouth)
* Anarthric

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Anterior Isometric Lingual Pressure Measured Using the TongueMeter Device | Participant will start using the tongue meter from day of enrollment. Baseline 1 : MAIP collected , Baseline 2: 5 weeks after baseline , then MAIP calculated at home , intensity of exercise set at 60% MAIP, 5 weeks of exercise at 60% MAIP
  Measurement Tool:
  Lingual pressure is measured using the TongueMeter, a handheld, pressure-sensing device designed to quantify tongue strength during isometric tasks. A calibrated intraoral pressure sensor is positioned against the hard palate. Participants are instructed to press the tongue upward with maximal effort for a standardized duration, and the device records the resulting pressure output.
  Unit of Measure:
  Lingual strength is quantified as peak pressure, reported in kilopascals (kPa).
  Outcome Variable:
  The primary outcome is the maximum peak lingual pressure (kPa) achieved across trials, with higher values indicating greater lingual strength
Videofluoroscopic Swallow Study | Baseline, Visit 1 (week 1), and Final Visit (week 10)swallowing safety/efficiency via DIGEST and PAS scores
  This measure assesses swallowing safety and efficiency in participants using standardized VFSS trials. Safety is quantified using the Penetration-Aspiration Scale (PAS) to capture airway compromise, while swallowing efficiency is measured with the Dynamic Imaging Grade of Swallowing Toxicity (DIGEST), which integrates residue severity and functional impact.
  Unit of Measure:
  PAS score for each swallow (ordinal 1-8)
  DIGEST grade for overall swallowing function (ordinal 0-4)
  Outcome Variable:
  The primary outcome is the frequency and severity of airway compromise (PAS) and overall dysphagia severity (DIGEST) during VFSS. Higher PAS and DIGEST scores indicate worse swallowing safety and efficiency.

SECONDARY OUTCOMES:
EAT-10 | From enrollment to the end of treatment at 10 weeks.
  The Eating Assessment Tool-10 (EAT-10) is a self-administered questionnaire used to screen for swallowing difficulties (dysphagia). It consists of 10 items that ask patients to rate symptoms such as effort during swallowing, coughing, and the impact of swallowing problems on quality of life. Each item is scored from 0 (no problem) to 4 (severe problem), with a total score of 3 or higher indicating possible dysphagia. It is quick, reliable, and widely used in both clinical and research settings.
Test of Mastication and Swallowing Solids | From enrollment to the end of treatment at 10 weeks.
  The Test of Masticating and Swallowing Solids (TOMASS) is a clinical assessment tool used to evaluate solid food swallowing efficiency. During the test, a patient is asked to eat a standardized cracker as quickly and safely as possible while the clinician records the number of bites, chews, swallows, and the total time taken. These measures provide insight into the efficiency and safety of oral intake. TOMASS is simple, non-invasive, and useful for identifying swallowing difficulties in both clinical practice and research.
ALS Functional Rating Scale | From enrollment to the end of treatment at 10 weeks.
  The ALS Functional Rating Scale (ALSFRS) is a standardized tool used to measure the functional status of individuals with amyotrophic lateral sclerosis (ALS). It assesses daily activities across key domains such as speech, swallowing, mobility, and respiratory function. Each item is scored from 0 (unable) to 4 (normal ability), with higher total scores indicating better functional status. The ALSFRS is widely used in both clinical care and research to track disease progression and treatment outcomes.
The Eating Tool Burden Questionnaire | To be given during at week 5 (baseline 2) and week 10 (final)
  The Eating Tool Burden Questionnaire (ETBQ) is a patient-reported outcome measure designed to evaluate the burden of eating and swallowing difficulties. It captures the physical, emotional, and social challenges patients experience during mealtimes. Responses are scored to reflect the severity of perceived burden, with higher scores indicating greater impact on daily life. The ETBQ is useful for understanding patient perspectives, guiding clinical care, and measuring changes over time in both practice and research.
Temporal Variability of Oral Diadochokinesis | From enrollment to the end of treatment at 10 weeks.
  Temporal Variability of Oral Diadochokinesis (DDK) is a measure used to assess the consistency and timing of rapid, repetitive speech movements, such as saying "pa," "ta," or "ka." It evaluates how evenly and steadily a person can produce these syllables, providing insight into motor speech control. Increased variability often indicates impaired oral motor coordination, which is common in neurological conditions like ALS. This measure is valuable in both clinical and research settings for monitoring speech function and disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Tabor Gray, Ph.D., Principal Investigator — Neuroscience Institute, Cathy J. Husman ALS Center

IPD SHARING:
Plan to Share IPD: Yes
Data will be disseminated in open access publication.
Supporting Information: Study Protocol
Time Frame: Data will be disseminated in open access publication.
Access Criteria: Data will be disseminated in open access publication.

DOCUMENTS (1):
  • Informed Consent Form (2025-08-14): https://cdn.clinicaltrials.gov/large-docs/90/NCT07295990/ICF_000.pdf